CLINICAL TRIAL: NCT05492734
Title: A Phase 1 Study to Assess the Feasibility of Non-invasive Dried Blood Sampling for Assessment of EDG-5506 Concentrations
Brief Title: A Study to Assess the Feasibility of Non-invasive Dried Blood Sampling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-5506-104
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Muscular Dystrophies
Keywords: Healthy Volunteers
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Drug: EDG-5506
  Interventions: Drug: EDG-5506

INTERVENTIONS:
Drug: EDG-5506 — single oral dose

SUMMARY:
This is a Phase I, open-label, single-dose, 1-period study to compare EDG-5506 concentrations measured from venous and capillary blood sampling in healthy adult subjects.

EDG-5506 is an investigational product designed to selectively modulate a fast skeletal muscle motor protein called myosin that is part of the contraction machinery of the damage-prone muscle fibers.

DETAILED DESCRIPTION:
Ten (10) healthy, adult male and female (of non-childbearing potential only) participants will be enrolled in the single-site study. Participants will receive a single oral dose of EDG-5506 on Day 1. Serial blood sampling will be collected pre-dose and up to 26 hours post-dose using venous blood sampling by venipuncture and capillary blood sampling by a capillary blood self-sampling device. On Day 3, participants will self-collect a capillary blood sample at home. The final on-site visit will be on Day 7 when a last blood sample will be collected using venous blood sampling by venipuncture and capillary blood sampling by a capillary blood self-sampling device.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, males or females, aged 19-55 years (inclusive) at the Screening visit.
2. Females must be of non-childbearing potential. Males with female partners must use a medically accepted contraceptive regimen or abstain from sexual intercourse for 90 days after dosing.
3. Non-smoker and must not have used any tobacco products within 3 months prior to the Screening visit.
4. Body weight greater than 50 kg and body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive at the Screening visit.
5. Medically healthy with no clinically significant findings for oculofacial and proximal limb strength assessments and swallowing function assessment, medical history, physical examination, laboratory profiles, vital signs, and ECGs.

Exclusion Criteria:

1. History of, or physical examination findings indicating clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases that, in the opinion of the PI, would render the subject being unsuitable for the study.
2. Female participants with a positive pregnancy test at the screening visit or are lactating.
3. Poor venous access and/or cannot tolerate venipuncture.
4. Unable to refrain from or anticipates the use of any drugs (including prescription and non-prescription medications, herbal remedies, vitamin supplements, or grapefruit/Seville orange containing products) beginning 14 days prior to dosing. Any drugs known to be moderate or strong inducers of CYP3A4 enzymes cannot be used within 28 days prior to dosing.
5. Participation in any other investigational drug study within 30 days prior to dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Difference in area under the concentration-time curve (AUC0-24, AUC0-26, AUC0-144 and AUC0-t) measurements for EDG-5506 in blood collected by capillary blood self-sampling versus venous blood sampling | 7 days
Plasma maximum measured drug concentration (Cmax) measurements for EDG-5506 in blood collected by capillary blood self-sampling versus venous blood sampling | 7 days
Time of maximum concentration (Tmax) measurements for EDG-5506 in blood collected by capillary blood self-sampling versus venous blood sampling | 7 days

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC0-24, AUC0-26, AUC0-144 and AUC0-t) measurements for EDG-5506 in plasma. | 7 days
Plasma maximum measured drug concentration (Cmax) measurements for EDG-5506 in plasma. | 7 days
Time of maximum concentration (Tmax) measurements for EDG-5506 in plasma. | 7 days
Incidence of treatment-emergent adverse events | 7 days
Incidence of abnormal clinical laboratory test results | 7 days
Incidence of abnormal vital signs | 7 days
Incidence of abnormal electrocardiograms (ECGs) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Sam Collins, MBBS, PhD, Study Chair — Edgewise Therapeutics, Inc.
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.edgewisetx.com